CLINICAL TRIAL: NCT04238299
Title: Application of Functional Renal MRI to Improve Assessment of Chronic Kidney Disease
Acronym: AFiRM
Status: Recruiting | Type: Observational
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Collaborators: University of Nottingham (Other); Queen Elizabeth University Hospital Glasgow (Unknown); Royal Infirmary of Edinburgh (Other); University of Edinburgh (Other); Newcastle University (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); University of Leeds (Other); The Leeds Teaching Hospitals NHS Trust (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other); University of Sheffield (Other); Northern Care Alliance NHS Foundation Trust (Other); University College, London (Other); University of Cambridge (Other); Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: DHRD/2018/100; 271043 (Other: IRAS)
Record Dates: First submitted 2020-01-20; First posted 2020-01-23 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stored samples: plasma, serum, urine and DNA at study entry Multiparametric renal MRI measures at study entry and after 2 years of follow up
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main study cohort: Patients with CKD recruited from specialist nephrology clinics
  Interventions: Diagnostic Test: Multiparametric renal MRI

INTERVENTIONS:
Diagnostic Test: Multiparametric renal MRI — Localiser scans; Kidney volume; Longitudinal (T1) relaxation time mapping; Diffusion weighted imaging (DWI); Phase Contrast MRI; Arterial spin labelling (ASL); Blood Oxygen Level Dependent (BOLD) mapping

SUMMARY:
Research question: Can multiparametric renal Magnetic Resonance Imaging (MRI) provide structural and functional assessment of the kidneys to deliver prognostic information and guide treatment options in chronic kidney disease (CKD)?

Aims and objectives:

1. To establish a multiparametric renal MRI protocol in CKD cohorts.
2. To use multiparametric MRI to characterise people with and without CKD progression.
3. To compare multiparametric renal MRI with 'gold-standard' renal biopsy to determine pathological processes of CKD progression that are detectable by MRI.

DETAILED DESCRIPTION:
The study will have three stages.

Stage 1: 45 people with CKD from nine UKRIN centres will undergo multiparametric MRI to test patient tolerance, data completeness and central data collection processes.

Stage 2: A multicentre, prospective cohort study of 450 people with CKD, collecting multiparametric renal MRI at baseline and 2 years. Long-term outcomes will be determined with efficient tracking of kidney failure events via the UK Renal Registry at 5 and 10 years.

Stage 3: A mechanistic sub-study of 45 patients (from Stage 2) who have had a routine renal biopsy. Detailed comparisons will be made between multiparametric MRI and histopathological changes. Tissue blocks will undergo quantitative analysis of fibrosis, capillary density and inflammation using immunohistochemistry techniques.

ELIGIBILITY:
Inclusion Criteria

* Age 18-75 years
* CKD category G3-4 or CKD category G1-2 with overt albuminuria (urine ACR>30mg/mmol)
* Capable of giving informed consent

Exclusion Criteria

* Autosomal dominant polycystic kidney disease (ADPKD)
* Glomerulonephritis (GN) actively receiving immunosuppression, or within the preceding 90 days.
* Multiple myeloma (MM)
* Acute Kidney Injury (AKI) within the preceding 90 days
* Solid organ transplant
* Known single kidney
* Contraindications to MRI (e.g. permanent pacemaker, metallic foreign bodies, claustrophobia etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic kidney disease
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2033-02-28 (Estimated)

PRIMARY OUTCOMES:
CKD progression | 10 years
  kidney failure (doubling of serum creatinine, eGFR<15ml/min or RRT) OR a 40% decline in eGFR

SECONDARY OUTCOMES:
Kidney failure events | 10 years
  Doubling of serum creatinine, eGFR<15ml/min or RRT
40% decline in eGFR from baseline | 10 years
eGFR trajectory | 2 years
  (ml/min/yr)
AKI events | 4 years
  AKI as per KDIGO serum creatinine criteria
Cardiovascular events | 4 years
All cause mortality | 10 years

OTHER OUTCOMES:
Renal MRI measures | 2 years
  As detailed in interventions section
Renal histology measures | Baseline
  Glomerulosclerosis score, extent of interstitial fibrosis, inflammation, peritubular capillary density, collagen accumulation, inflammatory cell subtypes

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Derby Hospital, Derby, Derbyshire, United Kingdom

REFERENCES:
- See also: Derby Clinical Trials Support Unit — https://www.uhdb.nhs.uk/derby-ctu